CLINICAL TRIAL: NCT00903890
Title: Cardiac Effects in Long-Term Survivors of Hodgkin's and Non-Hodgkin's Lymphoma After Radiation Therapy/Anthracycline Chemotherapy
Brief Title: Cardiac Effects in Long-Term Survivors of Hodgkin's and Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Louis Constine, Professor, University of Rochester
Other Study IDs: ULYM07056
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Individuals who have previously received radiation therapy and anthracycline chemotherapy for their Hodgkin's or non-Hodgkin's lymphoma.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey asking questions regarding the subjects cardiac and general health.

SUMMARY:
This study is to inquire by mailed survey regarding the cardiac and general health of patients previously treated for Hodgkin's and non-Hodgkin's lymphoma with radiation therapy/anthracycline chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Hodgkin's Lymphoma and Non Hodgkin's lymphoma who underwent Radiation Therapy (RT) to either a mantle or modified mantle field with or without adriamycin at the Wilmot Cancer Center at the University of Rochester are eligible for the study.

Exclusion Criteria:

* Any severe preexisting cardiac disease (e.g., arrhythmia, angina, coronary disease, myocardial infarction, or congestive heart failure) prior to diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated at the University of Rochester Department of Radiation Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2018-11 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Measure changes in Cardiac ejection fraction score | Post Radiation Treatment
Measure changes in perfusion imaging score on the radionuclide cardiac profusion scan | Post Radiation

CONTACTS AND LOCATIONS:
Overall Officials: Louis S Constine, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No